CLINICAL TRIAL: NCT04687618
Title: A Randomized Control Trial of Oxygen Assist Module in Preterm Infants on High Flow Nasal Cannula Support (ROAM)
Brief Title: Oxygen Assist Module in Preterm Infants on High Flow Nasal Cannula Support.
Acronym: ROAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Collaborators: Vapotherm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 291497
Record Dates: First submitted 2020-11-01; First posted 2020-12-29 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Preterm Birth
Keywords: Preterm; High Flow Nasal Cannula
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automatic control of FiO2 (Experimental): Infants randomized to this arm will be monitored using automatic oxygen control system on the High Flow Nasal Cannula. When infants oxygen saturation are out of the target range the OAM module on HFNC will adjust the oxygen delivery depending on the saturation of the infant to bring the saturation in the target range.
  Interventions: Device: High Flow Nasal Cannula withAutomatic control of FiO2 using OAM
- Manual Control of FiO2 (Active Comparator): Infants randomized to this arm will be receive oxygen delivery adjustments manually by the nursing and medical team taking care of the infants. When the infants oxygen saturation are out of the target range, the staff will manually adjust the oxygen delivery.
  Interventions: Device: High Flow Nasal Cannula with manual control of FiO2

INTERVENTIONS:
Device: High Flow Nasal Cannula withAutomatic control of FiO2 using OAM — The target oxygen saturation (SpO2) value will to be determined and set by the clinician according to specific patient needs. The target SpO2 in preterm infants is 90-95% with alarm limits at 89-96%. In automatic control of oxygen, the OAM automatically increases or decreases the FiO2 (oxygen delivery) setting on the Vapotherm Precision Flow based on pulse oximetry readings of the OAM. The target saturation will be set at 93% and the FiO2 will be adjusted by OAM to maintain the target saturation. The automated FiO2 setting can be overridden for a clinician pre-set period of time (30-120 sec) by simply manually adjusting the FiO2 on the Precision Flow. Automated control resumes after the clinicians pre-set period of time (30-120 sec) based on the current SpO2 and FiO2. The OAM utilizes a feedback control algorithm that receives a patient's oxygen saturation value from a build in pulse oximetry device (Masimo SET OEM - normal sensitivity, averaging time window set at 8 seconds).
  Arms: Automatic control of FiO2
Device: High Flow Nasal Cannula with manual control of FiO2 — In manual control of oxygen all FiO2 adjustments will be done by the clinical staff to maintain saturations between 90-95%. The alarm limits will be 89-96%.
  Arms: Manual Control of FiO2

SUMMARY:
Oxygen treatment is common in babies born early (preterm) and requiring intensive care. Having too much or too little oxygen can increase the risk of damage to the eyes and lungs, and contribute to death or disability. Preterm infants because of their immaturity experience episodes of low oxygen levels. The low oxygen episodes are primarily due to pauses in their breathing (Apnoea of prematurity) and immaturity of their lung. These episodes persist for weeks to months. The lower the gestation at birth the longer the duration of these events. Studies have shown that these episodes of low oxygen saturations especially if frequent and prolonged is associated with poor developmental outcome, severe eye disease and lung disease.

Traditionally, the oxygen delivery is manually adjusted when infant has low oxygen saturation. However previous studies have shown despite the best efforts the oxygen level can only be maintained less than half of the time and nearly a one-fifth of the time infant spends in low oxygen levels and nearly one-third of the time in high oxygen levels. With advancement in the neonatal care, preterm infants tend to spend more time on non invasive respiratory support. Now it is possible to maintain oxygen level in target range by using automatic control of oxygen delivery on non invasive support. With the proposed study, we would like to study the efficacy of automatic control of oxygen delivery in reducing the time spent in very low and high oxygen levels when infants are on non invasive respiratory support namely High Flow Nasal Cannula support.

DETAILED DESCRIPTION:
Supplemental oxygen remains by far the most commonly used 'drug' in neonatal intensive care units. The goal of oxygen therapy is to maintain normal oxygenation while minimizing hypoxemia and hypoxemia. Preterm infants are particularly vulnerable to oxygen toxicity and oxidative stress leading to retinopathy of prematurity (ROP), bronchopulmonary dysplasia (BPD), and periventricular leukomalacia (PVL). It's also well known that preterm infants experience hypoxic events which are primarily linked to cardiovascular instability and apnea of prematurity. These events vary as the infant matures. Martin R et al showed in their study that these hypoxic events peaked around 2-4 weeks and decreases by 6-8 weeks in preterm infants . Exposure to prolonged and frequent hypoxemic episodes has been associated with increased morbidity and mortality . Prolonged hypoxic events (Saturation less than 80% for more than 1 minute) have been associated with severe ROP and impaired neurodevelopmental outcome in survivors . Very high oxygen levels are equally harmful.

Peripheral oxygen saturation monitoring is standard of care in infants admitted to neonatal unit. Traditionally oxygen saturation (SpO2) targeting is carried out by manual adjustment of fraction of inspired oxygen (FiO2) by the caregiver based on the monitored oxygen saturation. However, in practice this is only partially achieved during routine care[6]. Hagadorn et al conducted a study in 14 centers and showed that preterm infants under 28 weeks' gestation receiving oxygen spent on average only 48% of the time with SpO2 within the prescribed target range, about 36% of the time above and 16% of the time with SpO2 below the target range.

Preterm infants have frequent fluctuations in SpO2 due to their cardio-respiratory instability requiring frequent adjustments of FiO2 . Consequently, these particularly vulnerable infants spend significant time with SpO2 outside intended range and are often exposed to extremes of hypoxemia and hyperoxaemia. The automatic oxygen control system continuously monitors the oxygen saturation and adjusts the oxygen delivery to maintain oxygen saturation within the target range. The safety, feasibility and efficacy of this mode of oxygen control have already been established. Automated control of FiO2 significantly improves compliance of oxygen saturation targeting and significantly reduces exposure to hypoxemia as well as hyperoxaemia. Automatic control of oxygen delivery is available in both invasive and non-invasive mode of ventilation. The HFNC Therapy is a common mode of non-invasive respiratory support in preterm infants. Oxygen Assist Module (OAM) is a system of automatic oxygen control available in the HFNC (Vapotherm Precision Flow).

Previous study looking at the efficacy of automated oxygen control with HFNC support mostly have been a crossover model and the study duration less than 48 hours . As previously mentioned, preterm infants experience hypoxic events for few weeks before cardiopulmonary maturation is established. Hence, it's important to study these events over a longer period of time. The objective of this randomized control trial is to evaluate the efficacy of OAM (Automatic oxygen Control) in reducing the extremes of oxygen saturations in preterm infants (<80% and >98%) through the entire period of HFNC respiratory support.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants {born at a gestation <33 weeks (23+0 to 32+6 weeks) }
* Receiving HFNC as respiratory support anytime during their stay in the neonatal support

Exclusion Criteria:

* Preterm infants more than equal to 33 weeks.
* Preterm infants with major congenital or chromosomal anomalies

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of time spent in extreme saturation (<80% and >98%) in preterm infants receiving HFNC as respiratory support. | Through study completion on an average of 3 months
  The primary outcome of this study is proportion of time spent in extreme saturation (<80% and >98%) in preterm infants receiving HFNC as respiratory support.

SECONDARY OUTCOMES:
Proportion of time spent in target saturation | Through study completion on an average of 3 months
  Proportion of time spent in target saturation
Proportion of time spent in saturation >95% | Through the study completion on an average of 3 months
  Proportion of time spent in saturation >95%
episodes of prolonged hypoxemia (SpO2 < 80% for more than 60 sec) | Through study completion on an average of 3 months
  episodes of prolonged hypoxemia (SpO2 < 80% for more than 60 sec)

CONTACTS AND LOCATIONS:
Overall Officials: Vrinda Nair, Principal Investigator — South Tees NHS Trust
Locations (1):
- James Cook University Hospital, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stoll BJ, Hansen NI, Bell EF, Shankaran S, Laptook AR, Walsh MC, Hale EC, Newman NS, Schibler K, Carlo WA, Kennedy KA, Poindexter BB, Finer NN, Ehrenkranz RA, Duara S, Sanchez PJ, O'Shea TM, Goldberg RN, Van Meurs KP, Faix RG, Phelps DL, Frantz ID 3rd, Watterberg KL, Saha S, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal outcomes of extremely preterm infants from the NICHD Neonatal Research Network. Pediatrics. 2010 Sep;126(3):443-56. doi: 10.1542/peds.2009-2959. Epub 2010 Aug 23. PMID 20732945
- [Background] Martin RJ, Wang K, Koroglu O, Di Fiore J, Kc P. Intermittent hypoxic episodes in preterm infants: do they matter? Neonatology. 2011;100(3):303-10. doi: 10.1159/000329922. Epub 2011 Oct 3. PMID 21986336
- [Background] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Carlo WA, Finer NN, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Schibler K, Newman NS, Ambalavanan N, Frantz ID 3rd, Piazza AJ, Sanchez PJ, Morris BH, Laroia N, Phelps DL, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Ehrenkranz RA, Watterberg KL, Higgins RD. Target ranges of oxygen saturation in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1959-69. doi: 10.1056/NEJMoa0911781. Epub 2010 May 16. PMID 20472937
- [Background] Reynolds PR, Miller TL, Volakis LI, Holland N, Dungan GC, Roehr CC, Ives K. Randomised cross-over study of automated oxygen control for preterm infants receiving nasal high flow. Arch Dis Child Fetal Neonatal Ed. 2019 Jul;104(4):F366-F371. doi: 10.1136/archdischild-2018-315342. Epub 2018 Nov 21. PMID 30464005
- [Background] Lal M, Tin W, Sinha S. Automated control of inspired oxygen in ventilated preterm infants: crossover physiological study. Acta Paediatr. 2015 Nov;104(11):1084-9. doi: 10.1111/apa.13137. PMID 26194933
- [Derived] Nair V, Kannan Loganathan P, Lal MK, Bachman TE, Fantl R. Randomised control trial of oxygen assist module in preterm infants on high-flow nasal cannula support. Arch Dis Child Fetal Neonatal Ed. 2023 Dec 15;109(1):65-69. doi: 10.1136/archdischild-2023-325661. PMID 37451840